CLINICAL TRIAL: NCT05851599
Title: Dose-ranging Study of Labisia Pumila Standardized Extract (SKF7®) for Obesity: a Randomized, Double-blind, Placebo-controlled, Phase-2 Study
Brief Title: Dose-Ranging Study of SKF7® for Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medika Natura Sdn Bhd (Industry)
Collaborators: Zach Biotech Depot Sdn Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSU-P-1-1019
Record Dates: First submitted 2023-01-31; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SKF7® - 375 mg (Experimental): Patients who meet the entry criteria for the study will be randomized to receive 375 mg SKF7® for 16 weeks
  Interventions: Other: SKF7® Labisia pumila standardized extract
- SKF7® - 562.5 mg (Experimental): Patients who meet the entry criteria for the study will be randomized to receive 562.5 mg SKF7® for 16 weeks
  Interventions: Other: SKF7® Labisia pumila standardized extract
- SKF7® - 750 mg (Experimental): Patients who meet the entry criteria for the study will be randomised to receive 750 mg SKF7® for 16 weeks
  Interventions: Other: SKF7® Labisia pumila standardized extract
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: SKF7® Labisia pumila standardized extract

INTERVENTIONS:
Other: SKF7® Labisia pumila standardized extract — Botanical extract of Labisia pumila (Kacip Fatimah)
  Other Names: SKF7®

SUMMARY:
This study has been designed as a randomized, double blinded, multi-centric, placebo controlled and phase II dose-ranging study. One group will receive placebo alone and the other three groups will receive IP twice daily (different dosages) for four months.

DETAILED DESCRIPTION:
Labisia pumila or Kacip Fatimah, a native Malaysian plant, has been used as traditional medicine for over 400 years by both men and women for multiple treatments. Studies in animal models showed that Labisia pumila extract could regulate body weight gain and visceral fat reduction. SKF7® is a standardized extract of Labisia pumila (Kacip Fatimah) from the Myrsinaceae family.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18 - 60 years.
2. Women aged 18 until before menopause.
3. BMI 30 - 37 kg/m2.
4. Waist circumference ≥ 60% of height.
5. Generally healthy or in the presence of co-morbidities of treated or untreated hypertension, diabetes or hyperlipidaemia.
6. Normotension or well-controlled mild hypertension (< 140/90 mmHg) with stable dosage of not more than 2 class drug combination (except beta blocker and diuretic) for at least 1 month.
7. Normoglycemic or non-insulin dependent diabetes mellitus (HbA1c ≤ 8.5%) with stable dosage of not more than 2 class drug combination (except sulphonylureas, TZDs and SGLT2 inhibitors) for at least 1 month.
8. Normolipidaemia or hyperlipidaemia (LDL ≤ 4.1 mmol/L and TG ≤ 5.6 mmol/L) with stable dosage of not more than 2 class drug combination for at least 1 month.
9. Agreed to maintain their current lifestyles (no changes in their diet and physical exercise) during the clinical trial period.
10. Willing to participate in the study by signing the informed consent.
11. Ability to provide written informed consent.

Exclusion Criteria:

1. Known hypersensitivity to any herbal product.
2. Known history of allergic reaction to microcrystalline cellulose, maltodextrin, tricalcium phosphate, silicon dioxide and glyceryl monostearate.
3. Pregnant or lactating women.
4. Taking any other weight loss therapy or who have lost more than 10% of their body weight within the last 6 months.
5. Taking regular herbal drugs or any supplements unless subjects willing to stop during the study.
6. Known HIV subjects.
7. Severe liver function impairment (ALT & AST > 3x ULN (upper limit of normal)
8. Renal function impairment (serum creatinine > 132.6 µmol/L)
9. Participating in other interventional clinical study or have taken other investigational drug within 30 days prior to screening.
10. Having endocrine disease that may affect weight such as hypothyroidism or Cushing's syndrome (by anamnesis).
11. Taking hormonal contraceptive within the last 3 months or planning to use it during the study.
12. Female patient of childbearing potential who is planning to get pregnant/male patient who is planning to have a child or do not agree to use non-hormonal contraception for the entire duration of the study.
13. Having heart diseases (e.g. heart failure, angina pectoris, or myocardial infarction), respiratory diseases (e.g. asthma or obstructive pulmonary disease), stroke, or ischemic heart failure.
14. Having malignant tumors within the last 5 years.
15. Participants who have narrow-angle glaucoma.
16. Participants who have cholelithiasis.
17. Participants with a neurologically or psychologically significant history of disease or who are currently suffering from the disease (e.g. schizophrenia, epilepsy, alcoholism, drug addiction, anorexia, hyperphagia, etc.).
18. Participants who have taken oral steroids (e.g. prednisone or its equivalent) within the last 3 months that may affect weight.
19. Participants who have taken b-blocker or diuretic drugs for hypertension, anorexiants, laxatives, thyroid hormone, amphetamine, cyproheptadine, phenothiazine, contraceptive or female hormones within the last 3 months that may affect weight.
20. Participants who have taken other treatments (e.g. insulin, blood thinning, antidepressants, selective serotonin reuptake inhibitors (SSRIs), barbiturate, antipsychotics, antiepileptic, or drugs concerned with abuse) within the last 5 years.
21. Participants who have anatomical condition or underwent anatomical changes which make it difficult/unable to conduct physical measurements.
22. Participants who underwent surgeries for weight reduction (e.g., gastroplasty or gastrectomy).
23. Participants who are judged as unable to comply with the study according to the findings of the clinical investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving more than or equal to 5% weight loss OR | Baseline Day 1 to Week 16
  Percentage of patients achieving more than or equal to 5% weight loss for SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo
Percentage of patients achieving more than or equal to 5 cm waist circumference reduction | Baseline Day 1 to Week 16
  Percentage of patients achieving more than or equal to 5 cm waist circumference reduction for SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo

SECONDARY OUTCOMES:
Percentage change from baseline in body weight (kg) at week 16 | Baseline Day 1 to Week 16
  SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo
Percentage change from baseline in waist circumference (cm) at week 16 | Baseline Day 1 to Week 16
  SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo
Percentage change from baseline in waist to height ratio at week 16 | Baseline Day 1 to Week 16
  SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo
Percentage change from baseline in BMI at week 16 | Baseline Day 1 to Week 16
  SKF7® (375 mg, 562.5 mg and 750 mg) versus placebo
Change in blood lipid concentrations. | Baseline Day 1 to Week 16
  The change in blood lipid concentrations (total cholesterol, triglyceride, HDL & LDL)
Incidence of AEs, SAEs and AEs leading to early discontinuation | Up to Follow up visit Up to Week 17
  Incidence of AEs, SAEs and AEs leading to early discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Vijayasingham, MBBS, MRCPS, Principal Investigator — Hospital Melaka, Malaysia
Locations (6):
- Malaysia (6):
  - Klinik Kesihatan Greentown, Ipoh
  - Klinik Kesihatan Kuang, Kuang
  - Hospital Melaka, Malacca
  - Klinik Kesihatan Masjid Tanah, Malacca
  - Hospital Tuanku Jaafar, Seremban
  - Klinik Kesihatan Seremban 2, Seremban

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swarna Nantha Y, Vijayasingham S, Adam NL, Vengadasalam P, Ismail M, Ali N, Chang LC, Ling LYL, Tee TT, Cheah YH. Labisia pumila standardized extract (SKF7(R)) reduces percentage of waist circumference and waist-to-height ratio in individuals with obesity. Diabetes Obes Metab. 2023 Nov;25(11):3298-3306. doi: 10.1111/dom.15229. Epub 2023 Aug 8. PMID 37551550